CLINICAL TRIAL: NCT06181422
Title: Comparative Study to Evaluate the Safety and Possible Efficacy of Metformin Versus Lactoferrin in ICU Patients With
Brief Title: Metformin and Lactoferrin in Sepsis in Icu
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Hemida, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: metformin and lactoferrin
Record Dates: First submitted 2023-12-04; First posted 2023-12-26 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Sepsis
Keywords: sepsis; metformin; lactoferrin
MeSH Terms: conditions — Sepsis | interventions — Metformin; Lactoferrin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1: Metformin (Active Comparator): Group1: (Metformin, n=30) who will receive metformin 500 mg three times daily.
  Interventions: Drug: Metformin
- Group 2 :Lactoferrin (Active Comparator): Group 2 :(Lactoferrin, n=30) who will receive lactoferrin 100 mg three times daily
  Interventions: Drug: Lactoferrin

INTERVENTIONS:
Drug: Metformin — metformin 500 mg
  Arms: Group1: Metformin
Drug: Lactoferrin — lactoferrin 100 mg
  Arms: Group 2 :Lactoferrin

SUMMARY:
Sepsis is a life-threatening organ dysfunction triggered by an unregulated response of a host to infection. Sepsis is a reason for substantial mortality and morbidity among intensive care unit (ICU) patients. 1 Therefore, the aim of our study is to compare the safety and efficacy of metformin and lactoferrin in ICU patients with sepsis.

DETAILED DESCRIPTION:
Sepsis is a life-threatening organ dysfunction triggered by an unregulated response of a host to infection. Sepsis is a reason for substantial mortality and morbidity among intensive care unit (ICU) patients. 1 The pathophysiology of sepsis has changed spectacularly over the last several decades. Significant comprehension into the components of the inflammatory response has been achieved. Inflammation contributes to endothelial injury and initiates coagulation pathways.2 The inflammatory reaction is mediated by the release of cytokines (tumor necrosis factor-alpha, interleukins, and prostaglandins) from neutrophils and macrophages. The cytokines trigger the extrinsic coagulation cascade and inhibit fibrinolysis. These overlapping processes end with organ dysfunction.3 The Sequential Organ Failure Assessment or SOFA score was developed to assess the acute morbidity of critical illness at a population level and has been extensively validated as a tool for this purpose across a range of healthcare settings and environments.4 Metformin is oral anti-diabetic agent that has positive effects such as antioxidant and anti-inflammatory properties which are considered potentially beneficial properties for management of septic patients. Previous studies showed that preadmission metformin use may reduce mortality in adult patients with sepsis and diabetes mellitus. Therefore, our study aims to test the potential efficacy of metformin in all subsets of patient with sepsis.5,6 Lactoferrin is a cationic glycoprotein and associated with many activities including the relevant anti-inflammatory one, especially associated to the downregulation of pro-inflammatory cytokines besides its anti-microbial and immunomodulatory effect.7 A previous study suggested that lactoferrin supplementation to enteral feeds with or without probiotics decreases late-onset sepsis in preterm infants without adverse effects and this encourage us to test its role in adult patients with sepsis.8 Therefore, the aim of our study is to compare the safety and efficacy of metformin and lactoferrin in ICU patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Age more than 18 years old.
  2. A diagnosis of sepsis according to the latest Sepsis definition.11
  3. Estimated GFR >45 ml/minute.

Exclusion Criteria:

Exclusion Criteria:

1. Pregnancy and breast feeding.
2. End stage hepatic disease.
3. End stage renal disease -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-06-09 (Estimated); Study Completion 2024-06-09 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is mortality rate | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Hemida, Principal Investigator — Tanta University
Locations (1):
- Tanta, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No